CLINICAL TRIAL: NCT04744207
Title: A Phase II, Randomized, Multi-center, Placebo-controlled, Double-blind Study to Investigate the Safety of GS-248, and Efficacy on Raynaud's Phenomenon (RP) and Peripheral Vascular Blood Flow, in Subjects With Systemic Sclerosis (SSc)
Brief Title: A Study to Investigate Safety of GS-248 and Efficacy on Raynauds' Phenomenon in Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gesynta Pharma AB (Industry)
Collaborators: Ergomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-2001
Record Dates: First submitted 2021-01-28; First posted 2021-02-08 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GS-248 (Experimental): GS-248, capsule, 120 mg, once daily for 4 weeks
  Interventions: Drug: GS-248
- Placebo (Placebo Comparator): placebo, capsule, once daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-248 — 120 mg, capsule, once daily for 4 weeks
  Arms: GS-248
Drug: Placebo — capsule, once daily for 4 weeks
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the safety, and evaluate the efficacy of GS-248 versus placebo on Raynaud's Phenomenon (RP) in subjects with Systemic Sclerosis (SSc).

DETAILED DESCRIPTION:
The primary objective of this study is to determine the safety, and evaluate the efficacy of GS-248 versus placebo on Raynaud's Phenomenon (RP) in subjects with Systemic Sclerosis (SSc).

This is a randomized, double-blind, placebo-controlled study conducted in multiple sites in 4 countries in Europe. Approximately 80 subjects will be randomized in a 1:1 allocation to receive either GS-248 (120 mg) or placebo once daily. The study will comprise an enrolment period, a treatment period, and a follow-up period, with a total of 5 study visits over approximately 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide signed and dated written informed consent before the conduct of any study-specific procedures.
* Male and female subjects aged 18-75 years inclusive.
* Systemic Sclerosis diagnosed according to European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) criteria (van den Hoogen F et al. 2013). Subjects with signs of other autoimmune diseases (e.g. Sjögren's syndrome, myositis, rheumatoid arthritis) could be included if SSc is the dominating phenotype.
* Raynaud attacks typically ≥7 times per week during the last 4 weeks prior to screening despite background medication (only allowed vasodilatory therapy is calcium channel blockers or PDE-5 inhibitors).
* Women of childbearing potential must be using a highly effective method of contraception to avoid pregnancy throughout the study and for 4 weeks after the last dose of Investigational Medicinal Product in such manner that the risk of pregnancy is minimised.
* Women must not be pregnant or breastfeeding.
* Male subjects to agree to use condom in combination with use of contraceptive methods with a failure rate of <1% to prevent pregnancy and drug exposure of a partner, and refrain from donating sperm from the first date of dosing until 3 months after last dosing of the IMP.
* Ability of subjects to participate fully in all aspects of this clinical trial.

Exclusion Criteria:

* Systemic Sclerosis disease duration of greater than 120 months from first non-Raynaud manifestation
* Current smokers or stopped smoking <3 months prior to Visit 1.
* Dose-change or initiation of vasodilating substances (calcium blockers or PDE-5 inhibitors) within 4 weeks prior to Visit 1.
* Use of iloprost or other intravenous (iv) or po prostacyclin receptor agonist within 4 weeks prior to Visit 1.
* Ongoing treatment with immunosuppressive therapies (other than mycophenolate) including, but not restricted to; cyclophosphamide, azathioprine, methotrexate, or cyclosporine, or use of those medications within 4 weeks of trial entry.
* Use of systemic corticosteroids during 4 weeks before screening and during the course of the study.
* Concurrent serious medical condition, with special attention to cardiovascular conditions, which in the opinion of the Investigator makes the subject not suitable for this study.
* Prolonged QTcF interval defined as a mean QTcF >450 msec.
* Creatinine clearance <50 mL/min (determined by Cockcroft-Gault equation) at Screening.
* Active digital ulcer (DU) within 4 weeks prior to Visit 1.
* Clinically meaningful laboratory abnormalities at Screening (Visit 1), as determined and documented by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Edenius, Study Director — Gesynta Pharma
Locations (12):
- Investigator site, Ghent, Belgium
- Investigator Site, Nijmegen, Netherlands
- Poland (3):
  - Investigator site, Gdansk
  - Investigator Site, Krakow
  - Investigator site, Lublin
- United Kingdom (7):
  - Investigator site, Bath
  - Investigator site, Cambridge
  - Investigator Site, Dundee
  - Investigator site, Leeds
  - Investigator Site, Liverpool
  - Investigator Site, London
  - Investigator site, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In addition to fulfilling all eligibility criteria, subjects must fulfil the following criteria to be randomised:
  •≥7 RP attacks during the last week of the run-in period as captured in the eDiary, with no more than 2 days without RP attacks.
  •Compliance with the eDiary during the 7 most recent days prior to baseline (Visit 2), excluding the visit day itself, defined as having submitted ≥5 days of eDiary records (out of a possible 7 days) for RCS and RP during that period.
Pre-assignment Details: The run-in period was 14-21 days prior to Day 1, Baseline visit (the first dose of IMP).
  Of the 94 subjects enrolled into the study 69 subjects met the eligiblity criteria for randomization after the run-in period and were assigned to a treatment group.
Groups:
- GS-248: Participants received GS-248, (supplied as 40 mg capsules) Each single dose consisted of 3 capsules constituting a total of 120 mg, once daily for 4 weeks
  GS-248: 120 mg, capsule, once daily for 4 weeks
- Placebo: Participants received placebo, (supplied as 3 capsules), once daily for 4 weeks
  Placebo: capsule, once daily for 4 weeks
Period: Treatment
Arm/Group | GS-248 | Placebo
Started | 33 | 36
Completed | 30 | 34
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 1 | 2
Period: Follow-up
Arm/Group | GS-248 | Placebo
Started | 30 | 34
Completed | 30 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GS-248 | Placebo | Total
Number analyzed (Participants) | 33 | 36 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 32 | 62
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (10.6) | 50.6 (10.6) | 49.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 33 | 60
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 34 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Netherlands | 2 | 3 | 5
  Belgium | 2 | 1 | 3
  Poland | 17 | 20 | 37
  United Kingdom | 12 | 12 | 24
Stratification factors FAS [Count of Participants; unit: Participants] — Background vasodilatory treatment
  Participants
    Ca-blockers | 18 | 19 | 37
    PDE-5 inhibitors | 9 | 10 | 19
    No treatment | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 4 in the Number of Raynaud Attacks Per Week.
Description: Patient reported number of Raynaud's attacks per day as registered in electronic diary.
Time Frame: From baseline to week 4, i.e. the 7 most recent days prior to Visit 2 and Visit 4 respectively
Measure: Least Squares Mean (95% Confidence Interval); unit: number of attacks
Arm/Group | GS-248 | Placebo
Number analyzed (Participants) | 33 | 36
number of attacks | -3.41 [-5.83 to -0.99] | -4.22 [-6.48 to -1.96]
Statistical Analysis 1: Comparison: GS-248 vs Placebo; Test type: Superiority; p < 0.05, ANCOVA; Least squares mean estimate = 0.81, 95% CI 2-sided [-2.48 to 4.10]

2. Secondary Outcome: Mean Change From Baseline to Week 4 in the Raynaud's Condition Score.
Description: Patients reported Raynaud's Condition Score (RCS) once a day in an electronic diary.
  RCS is a validated numeric rating scale (from 0 to 10) answering the question "What difficulty did you have today with your Raynaud's condition?" where a score of '0' = 'No difficulty', and a score of '10' = 'Extreme difficulty'.
Time Frame: From baseline to week 4, i.e. the 7 most recent days prior to Visit 2 and Visit 4 respectively
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | GS-248 | Placebo
Number analyzed (Participants) | 33 | 36
score | -0.99 [-1.54 to -0.45] | -0.95 [-1.45 to -0.46]

3. Secondary Outcome: Mean Change From Baseline to Week 4 in Pain Experienced During Raynaud Attacks.
Description: The patient reported the experienced pain of each Raynaud attack using a Numeric Rating Scale (NRS) from 0 to 10 in an electronic diary where '0'='No pain' and '10'='Worst imaginable pain'.
Time Frame: From baseline to week 4, i.e. the 7 most recent days prior to Visit 2 and Visit 4 respectively
Measure: Least Squares Mean (95% Confidence Interval); unit: numeric rating scale
Arm/Group | GS-248 | Placebo
Number analyzed (Participants) | 33 | 36
numeric rating scale | -0.65 [-1.16 to -0.14] | -0.60 [-1.07 to -0.13]

4. Secondary Outcome: Mean Change From Baseline to Week 4 in the Mean Duration of Raynaud's Attacks
Description: The patient reported the start time (hh:mm) and stop time (hh:mm) of each Raynaud's attack in the electronic diary.
Time Frame: From baseline to week 4, i.e. the 7 most recent days prior to Visit 2 and Visit 4 respectively
Measure: Least Squares Mean (95% Confidence Interval); unit: LN (minutes); back-transformed
Arm/Group | GS-248 | Placebo
Number analyzed (Participants) | 33 | 36
LN (minutes); back-transformed | 1.06 [0.87 to 1.29] | 0.89 [0.74 to 1.08]

5. Secondary Outcome: Mean Change From Baseline to Week 4 in the Cumulative Duration of Raynaud Attacks.
Description: The patient reported the start time (hh:mm) and stop time (hh:mm) of each Raynaud's attack in the electronic diary.
Time Frame: From baseline to week 4, i.e. the 7 most recent days prior to Visit 2 and Visit 4 respectively
Measure: Least Squares Mean (95% Confidence Interval); unit: LN (minutes); back-transformed
Arm/Group | GS-248 | Placebo
Number analyzed (Participants) | 33 | 36
LN (minutes); back-transformed | 0.70 [0.51 to 0.98] | 0.61 [0.45 to 0.82]

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected during the full study period from the signing of the ICF until the last study visit (2-3 weeks run-in period, 4 weeks treatment period and 2-3 weeks follow-up period; i.e. 8-10 weeks).
Arm/Group | GS-248 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 1/36
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/36
Other Adverse Events (participants affected / at risk) | 10/33 | 9/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GS-248 (N=33) | Placebo (N=36)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GS-248 (N=33) | Placebo (N=36)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 6 (18) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT04744207/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT04744207/SAP_001.pdf